CLINICAL TRIAL: NCT06809400
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY4006896 in Healthy Participants and Participants With Parkinson's Disease
Brief Title: A Study of LY4006896 in Healthy Participants and Participants With Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27270; J5V-MC-ORAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single-blind study where the participants, investigator, and site personnel (except pharmacy staff) are blinded to study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A LY4006896 + Placebo (Experimental): Healthy participants will receive a single escalating dose of LY4006896 and matching placebo.
  Interventions: Drug: LY4006896
- Part B LY4006896 + Placebo (Experimental): Participants with Parkinson's disease will receive multiple escalating doses of LY4006896 and matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4006896 — Administered intravenously (IV)
  Arms: Part A LY4006896 + Placebo
Drug: Placebo — Administered IV
  Arms: Part B LY4006896 + Placebo

SUMMARY:
The purpose of this study is to generate evidence of the safety, tolerability, and pharmacokinetics/pharmacodynamics of IV LY4006896 compared with placebo in healthy participants and participants with Parkinson's disease.

DETAILED DESCRIPTION:
The screening period will be up to 120 days for participants with Parkinson's disease who receive 4 doses, and up to 35 days for healthy participants who receive 1 dose. The treatment and follow-up duration will be up to 61 weeks for participants with Parkinson's disease, and 48 weeks for healthy participants. The total study duration will be up to 78 weeks for participants with Parkinson's disease, and 53 weeks for healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Part A Single Ascending Dose (SAD) and B Multiple Ascending Dose (MAD)

* Have a body mass index within the range of 18 to 34 kilogram/square meter (kg/m²) (inclusive).
* For Japanese participants: To qualify as a participant of first-generation Japanese origin, the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.
* Have venous access sufficient to allow for blood sampling or administration of study intervention for IV administration, or both.

Part A (SAD) Only

* Participant must be 30 to 85 years of age (inclusive), at the time of signing the informed consent
* Are overtly healthy
* For Chinese participants: To qualify as Chinese for this study, all 4 of the participant's biological grandparents must be exclusive Chinese descent and born in China.

Part B (MAD) Only

* Participant must be 40 to 85 years of age (inclusive), at the time of signing the informed consent
* Diagnosis of Parkinson's disease per United Kingdom (UK) Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria.
* If presently untreated for Parkinson's disease, clinical status is not expected to require changes in symptomatic treatment within 52 weeks from baseline.
* If presently being treated for Parkinson's disease, receiving a stable dose of symptomatic dopaminergic therapy, including monoamine oxidase-B inhibitor, levodopa/carbidopa or dopamine agonist for at least 90 days prior to baseline and not expected to change within 52 weeks.
* Have a Montreal Cognitive Assessment (MoCA) score of greater than or equal to (≥) 24.

Exclusion Criteria:

Part A (SAD) and B (MAD)

* Have significant neurological disease affecting the central nervous system (CNS) (other than Parkinson's disease in Part B cohorts) that may affect the participant's ability to complete the study.
* Have a history or presence of serious or unstable illnesses or conditions that, in the investigator's opinion, could interfere with the analyses in this study, or increase risk for study intervention administration, or result in a participant's life expectancy of less than 24 months.
* Have known allergies to LY4006896, related compounds, or any components of the formulation, or history of allergic reactions to any transferrin receptor antibodies.
* Have significant allergies to humanize monoclonal antibodies.
* Have clinically significant multiple or severe drug allergies (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis); or intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions.
* Have history or presence of uncontrolled asthma, significant autoimmune disease, hereditary angioedema, or known history of common variable immune deficiency.
* Evidence of clinically significant anemia.

Part A (SAD) Only

* Have an abnormal blood pressure or pulse rate, or both, as determined by the investigator, or a preexisting history of hypertension.

Part B (MAD) Only

* Have an abnormal blood pressure or pulse rate, or both, as determined by the investigator, or have uncontrolled hypertension, defined as a systolic blood pressure >150 mm Hg or a diastolic blood pressure >95 mm Hg at Screening or Treatment Visits.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Part A | Baseline to Week 48
Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) Part A | Baseline to Week 48
Number of Participants with One or More SAEs Part B | Baseline to Week 61
Number of Participants with One or More TEAEs Part B | Baseline to Week 61

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4006896 ARC-Associated Antisense Part A | Baseline to Week 48
PK: Cmax of LY4006896 ARC-Associated Antisense Part B | Baseline to Week 61
PK: Area Under the Concentration versus Time Curve (AUC) of LY4006896 ARC-Associated Antisense Part A | Baseline to Week 48
PK: AUC of LY4006896 ARC-Associated Antisense Part B | Baseline to Week 61
Effect of LY4006896 on Aggregation-Competent Alpha-Synuclein in Skin Part B | Baseline to Week 61
  Alpha-synuclein seed amplification positivity
Effect of LY4006896 on Aggregation-Competent Alpha-Synuclein in Cerebrospinal Fluid (CSF) Part B | Baseline to Week 61
  Alpha-synuclein seed amplification positivity

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (11):
  - Collaborative Neuroscience Network - CNS, Los Alamitos, California
  - K2 Medical Research, LLC, Maitland, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Charter Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - K2 Medical Research, LLC, The Villages, Florida
  - Charter Research, The Villages, Florida
  - QUEST Research Institute, Farmington Hills, Michigan
  - PPD Development, LP, Austin, Texas
  - Evergreen Health Research, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Japan (2):
  - P-One Clinic, Hachiōji
  - Oita University Hospital, Yufu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4006896 in Healthy Participants and Participants With Parkinson's Disease — https://trials.lilly.com/en-US/trial/584136